CLINICAL TRIAL: NCT02441803
Title: Allogeneic Hematopoietic Stem Cell Transplantation as Initial Salvage Therapy for Patients With Primary Induction Failure Acute Myeloid Leukemia Refractory to High-Dose Cytarabine-Based Induction Chemotherapy
Brief Title: Allogeneic Hematopoietic Stem Cell Transplantation (AlloSCT) Initial Salvage Therapy for Induction Failure Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0358; NCI-2015-00849 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-05-05; First posted 2015-05-12 (Estimated); Results first posted 2024-01-17 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Leukemia
Keywords: Leukemia; Acute myeloid leukemia; AML; Refractory; Allogeneic hematopoietic stem cell transplantation; AHSCT; Busulfan; Busulfex; Myleran; Fludarabine; Fludarabine Phosphate; Fludara; Clofarabine; Clofarex; Clolar; Total body irradiation; TBI; XRT; Thymoglobulin; ATG (Rabbit); Rabbit antithymocyte Globulin; Rabbit Antilymphocyte Globulin; Rabbit ATG; rATG; Stem cell infusion; Cyclophosphamide; Cytoxan; Neosar; Tacrolimus; Prograf; Mycophenolate mofetil; MMF; CellCept; Decitabine; Dacogen; Cytarabine; Ara-C; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride; Idarubicin; Idamycin
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — Busulfan; fludarabine; fludarabine phosphate; Clofarabine; Whole-Body Irradiation; thymoglobulin; Cyclophosphamide; Tacrolimus; Mycophenolic Acid; Decitabine; Cytarabine; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Matched Sibling Donor Group (Experimental): Salvage Chemotherapy Before Transplant: Decitabine 20 mg/m2 by vein on Days 1 - 5. Cytarabine 1 g/m2 by vein on Days 6 - 10. Idarubicin 10 mg/m2 by vein on Days 6 - 8. Clofarabine 15 mg/m2 by vein on Days 6 - 9.
  Stem Cell Transplant: Test dose Busulfan 32 mg/m2 by vein on Day -8. Busulfan AUC 5,000 by vein on Days -6 to -3. Fludarabine 10 mg/m2 by vein on Days -6 to -3. Clofarabine 40 mg/m2 by vein on Days -6 to -3. Stem cell infusion performed on Day 0.
  Interventions: Drug: Busulfan; Drug: Fludarabine; Drug: Clofarabine; Biological: Stem Cell Infusion; Drug: Decitabine; Drug: Cytarabine; Drug: Idarubicin
- Haploidentical Donor Group (Experimental): Salvage Chemotherapy Before Transplant: Decitabine 20 mg/m2 by vein on Days 1 - 5. Cytarabine 1 g/m2 by vein on Days 6 - 10. Idarubicin 10 mg/m2 by vein on Days 6 - 8. Clofarabine 15 mg/m2 by vein on Days 6 - 9.
  Stem Cell Transplant: Test dose Busulfan 32 mg/m2 given by vein on Day -8. Busulfan AUC 5,000 by vein on Days -6 to -3. Fludarabine 10 mg/m2 by vein on Days -6 to -3. Clofarabine 40 mg/m2 by vein on Days -6 to -3. Total body irradiation (TBI) delivered at 2Gy on Day -2. Stem cell infusion performed on Day 0. Cyclophosphamide 50 mg/kg by vein on Days +3 and +4. Tacrolimus 0.015 mg/kg/day by vein or mouth on Day +5. Mycophenolate mofetil 15 mg/kg/dose by vein or by mouth three times a day from Day +5 to Day+100.
  Interventions: Drug: Busulfan; Drug: Fludarabine; Drug: Clofarabine; Radiation: Total Body Irradiation (TBI); Biological: Stem Cell Infusion; Drug: Cyclophosphamide; Drug: Tacrolimus; Drug: Mycophenolate mofetil; Drug: Decitabine; Drug: Cytarabine; Drug: Idarubicin
- Matched Unrelated Donor Group (Experimental): Salvage Chemotherapy Before Transplant: Decitabine 20 mg/m2 by vein on Days 1 - 5. Cytarabine 1 g/m2 by vein on Days 6 - 10. Idarubicin 10 mg/m2 by vein on Days 6 - 8. Clofarabine 15 mg/m2 by vein on Days 6 - 9.
  Stem Cell Transplant: Test dose Busulfan 32 mg/m2 given by vein on Day -8. Busulfan AUC 5,000 by vein on Days -6 to -3. Fludarabine 10 mg/m2 by vein on Days -6 to -3. Clofarabine 40 mg/m2 by vein on Days -6 to -3. Thymoglobulin 2.0 mg/Kg by vein on Days -3 and -2. Stem cell infusion performed on Day 0.
  Interventions: Drug: Busulfan; Drug: Fludarabine; Drug: Clofarabine; Drug: Thymoglobulin; Biological: Stem Cell Infusion; Drug: Decitabine; Drug: Cytarabine; Drug: Idarubicin

INTERVENTIONS:
Drug: Busulfan — Test dose Busulfan 32 mg/m2 given by vein on Day -8. Busulfan AUC 5,000 by vein on Days -6 to -3.
  Other Names: Busulfex; Myleran
Drug: Fludarabine — Fludarabine 10 mg/m2 by vein on Days -6 to -3.
  Other Names: Fludarabine Phosphate; Fludara
Drug: Clofarabine — Salvage Chemotherapy Before Transplant: Clofarabine 15 mg/m2 by vein on Days 6 - 9.
  Stem Cell Transplant: Clofarabine 40 mg/m2 by vein on Days -6 to -3.
  Other Names: Clofarex; Clolar
Radiation: Total Body Irradiation (TBI) — Total body irradiation (TBI) delivered at 2Gy on Day -2.
  Other Names: TBI; XRT
  Arms: Haploidentical Donor Group
Drug: Thymoglobulin — Thymoglobulin 2.0 mg/Kg by vein on Days -3 and -2.
  Other Names: ATG (Rabbit); Rabbit Antithymocyte Globulin; Rabbit Antilymphocyte Globulin; Rabbit ATG; rATG
  Arms: Matched Unrelated Donor Group
Biological: Stem Cell Infusion — Fresh or cryopreserved bone marrow or peripheral blood (PB) progenitor cells infused on Day 0. Goal is to infuse 4 X 106 CD34+ cells/kg if PB or >3.0 X 108 marrow mononuclear cells/kg if bone marrow.
Drug: Cyclophosphamide — Cyclophosphamide 50 mg/kg by vein on Days +3 and +4.
  Other Names: Cytoxan; Neosar
  Arms: Haploidentical Donor Group
Drug: Tacrolimus — Tacrolimus 0.015 mg/kg/day by vein or mouth on Day +5.
  Other Names: Prograf
  Arms: Haploidentical Donor Group
Drug: Mycophenolate mofetil — Mycophenolate mofetil 15 mg/kg/dose by vein or by mouth three times a day from Day +5 to Day+100.
  Other Names: MMF; CellCept
  Arms: Haploidentical Donor Group
Drug: Decitabine — 20 mg/m2 by vein on Days 1 - 5.
  Other Names: Dacogen
Drug: Cytarabine — 1 g/m2 by vein on Days 6 - 10.
  Other Names: Ara-C; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride
Drug: Idarubicin — 10 mg/m2 by vein on Days 6 - 8.
  Other Names: Idamycin

SUMMARY:
Objectives:

Primary Objectives:

1. To determine the safety and feasibility of allogeneic hematopoietic stem cell transplantation (AHSCT) as initial salvage treatment for patients with primary induction failure (PIF) acute myeloid leukemia (AML).
2. To determine efficacy of AHSCT following decitabine, clofarabine, idarubicin, and cytarabine (DCIA) salvage chemotherapy evaluated by overall response rate (RR), defined as complete response (CR) or CR without platelet recovery (CRp) or CR with insufficient hematological recovery (CRi).

Secondary Objectives:

1. To determine the percentage of patients with PIF AML eligible for AHSCT after up to 2 courses of induction chemotherapy.
2. To determine the early treatment-related mortality (TRM) (within first 4 weeks of first salvage chemotherapy regimen with DCIA and day 100 TRM after AHSCT.
3. To determine the efficacy DCIA regimen as salvage chemotherapy for patients with PIF AML (% of patients who achieve </=5% bone marrow blasts prior to AHSCT.
4. To determine the TRM at 1 year, relapse rate (RR), overall survival (OS) and event-free survival (EFS) for patients with PIF AML treated with DCIA followed by early AHSCT.

DETAILED DESCRIPTION:
Salvage Chemotherapy Before Transplant:

Study Drug Administration:

On Days 1-5, you will receive decitabine 1 time each day by vein over about 1-3 hours.

On Days 6-10:

* You will receive cytarabine 1 time a day by vein over about 1-3 hours.
* On Days 6-8 only, you will receive idarubicin 1 time a day by vein over about 30 minutes.
* On Days 6-9 only, you will receive clofarabine 1 time a day by vein over about 1-2 hours.

Study Visits:

After your last study drug dose:

* Blood (about 2 teaspoons) will be drawn to check your kidney and liver function.
* You will have an echocardiogram (ECHO) or multigated acquisition (MUGA) scan to check your heart function.
* You will have a lung function test.

On Day 21 (+/- 7 days), you will have a bone marrow biopsy/aspirate to check the status of the disease. To collect a bone marrow biopsy/aspirate, an area of the hip is numbed with anesthetic, and a small amount of bone and bone marrow is withdrawn through a large needle.

If the results of your bone marrow biopsy/aspirate, blood tests, and heart and lung function tests show that you are eligible to receive an allogeneic stem cell transplant, you will be asked to sign a separate informed consent for the transplant.

If the results of your bone marrow aspirate/biopsy, blood tests, and heart and lung function tests show that you are not eligible to receive an allogeneic stem cell transplant you will not receive it. The study staff will call you and ask how you are feeling and about any other drugs you may be taking every 3 months for 2 years after your last study drug dose. These calls should last about 5 minutes each.

If you are found to NOT be eligible to receive an allogeneic stem cell transplant, your doctor will discuss other treatment options with you.

Stem Cell Transplant:

Study Drug Administration, Pharmacokinetic (PK) Testing, and Stem Cell Transplant:

For a stem cell transplant, the days before you receive your stem cells are called minus days. The day you receive the stem cells is called Day 0. The days after you receive the stem cells are called plus days.

You will receive a dose of busulfan by vein over about 45 minutes to 1 hour as an outpatient or as an inpatient on Day -8. With the first busulfan infusion, blood (about 1 teaspoon each time) will be drawn for pharmacokinetic (PK) testing about 11 times over 11 hours before and after you receive your first dose of busulfan. PK testing measures the amount of study drug in the body at different time points. The study staff will tell you the blood testing schedule. Test doses are used to study how your body breaks down busulfan and decide the dose of busulfan that you will receive on Days -6 through -3.

A heparin lock line will be placed in your vein before the PK testing to lower the number of needle sticks needed for these draws. If for any reason it is not possible for the PK tests to be performed, you will receive the standard dose of busulfan.

On Day -7, you will rest.

On Days -6 through -3, you will receive fludarabine by vein over 1 hour, clofarabine by vein over 1 hour, and then busulfan by vein over 3 hours.

On Days -3 and -2, if you will receive stem cells from a matched unrelated donor, you will receive ATG by vein over 4 hours each day.

On Day -2, if you will receive stem cells from a haploidentical donor, you will receive total body irradiation (TBI) one time. TBI involves the delivery of high doses of radiation designed to destroy cancer cells and/or lower the immune system in order to lower the risk of the body rejecting the new stem cells.

On Day -2, you will receive tacrolimus by vein over 24 hours every day until you are able to take it by mouth. Tacrolimus is designed to weaken the immune system and lower the risk of graft-versus-host-disease (GVHD - a reaction of the donor's immune cells against your body). After you are able to take tacrolimus by mouth, you will take it every day for about 6 months, or until the doctor thinks it is safe to stop.

On Day -1, you will rest. If you will receive stem cells from a matched sibling donor, you will rest on Days -2 and -1.

On Day 0, you will receive the donor's stem cells by vein. The infusion will last anywhere from about 30 minutes to several hours.

If you will receive stem cells from a haploidentical donor:

After the stem cell infusion, you will receive tacrolimus to help lower the risk of GVHD. Tacrolimus will be given by vein non-stop for about 2 weeks. After the 2 weeks of taking tacrolimus by vein, you will take tacrolimus by mouth as a pill for at least 4 months after the transplant.

On Days +3 and +4, you will receive cyclophosphamide by vein over 3 hours. Cyclophosphamide is given to lower the immune system in order to lower the risk of GVHD.

If you receive stem cells from a matched sibling or matched unrelated donor:

On Days +1, +3, +6, and +11, you will receive methotrexate by vein over 30 minutes. Methotrexate is given to help prevent GVHD.

Study Testing:

Before you are sent home from the hospital and/or clinic, you will receive additional written instructions. These instructions will include how often you will come to the hospital/clinic, which standard drugs you will take at home, and what side effects you may have and what to do for them.

After finishing the chemotherapy and transplant, your follow-up care will be routine standard of care follow-up that all patients receiving allogeneic stem cell transplantation receive. At each visit, you will have a physical exam. You will be asked about any side effects you may have had. Blood (about 1 tablespoon) will be drawn for routine tests. If the doctor thinks it is needed, you will have a bone marrow aspiration to check the status of the disease. To collect a bone marrow aspirate, an area of the hip or other site is numbed with anesthetic, and a small amount of bone marrow is withdrawn through a large needle.

Length of Treatment:

After 2 years, your participation in this study will be over. You may be taken off study early if the disease gets worse, if your transplant does not "take" (graft failure), if you are unable to follow study directions, if your doctor thinks it is in your best interest, if the study is stopped, or if you choose to leave the study early.

If for any reason you want to leave the study early, you must talk to the study doctor. It may be life-threatening to leave the study after you have started to receive the study drugs but before you receive the stem cell transplant because your blood cell counts will be dangerously low.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 18-60 years.
2. Patients with diagnosis of AML, judged primary refractory after up to 2 courses of AML induction therapy (> 5% blasts on day 21 (+/-7 days) bone marrow aspirate and/or biopsy from the beginning of induction chemotherapy, up to 42 days).
3. Eastern Cooperative Oncology Group (ECOG) Performance Status </= 2.
4. Adequate major organ function:, defined as: a) Serum creatinine </= 3 mg/dL; b) Total bilirubin </= 2.5 mg/dL; c) ALT (SGPT) </= 3 x ULN or </= 5 x ULN if related to disease; d) Cardiac ejection fraction >/= 40% (by either ECHO or MUGA).
5. Willingness to have an allogeneic transplant.
6. Patient or patient's legal representative able to provide written informed consent.
7. Patients are required to meet the following criteria to proceed to AHSCT:
8. Donor criteria: Availability of a donor either an HLA matched sibling donor (MSD) or a haploidentical (5-9/10 HLA matched); alternatively a 8/8 HLA matched unrelated donor (MUD) by high resolution typing is immediately available;
9. Disease criteria: Day 21 (+/-7 days) bone marrow aspiration or biopsy from the beginning of salvage DCIA: a. In complete morphologic remission with <5% bone marrow blasts, or b. Aplastic (<10% bone marrow cellularity), and cytopenic with an absolute neutrophil count (ANC) less than 1,000/µL, or c. Low disease burden with < 30% BM blasts, with recovery of peripheral blood (PB) WBC (ANC>1,000/µL) and <5% circulating blasts.
10. Adequate organ function criteria: a. Serum creatinine clearance >/= 50 ml/min (calculated by Cockcroft-Gault formula); b. Total bilirubin </= 2 times upper limit of normal (x ULN) (3 x ULN if considered to be due to leukemic involvement or Gilbert's syndrome); c. Alanine aminotransferase (ALT) </= 3 x ULN (5.0 x ULN if considered to be due to leukemic involvement); d. LVEF >/= 40% on ECHO or MUGA; e. DLCO >/= 50% predicted after correction for hemoglobin (must be performed in patients with history of smoking or lung disease;); DLCO may be omitted in patients without history of pulmonary disease if approved by the Study Chair.
11. No active infection: Patients should be afebrile. If present, pulmonary infiltrates or other sites of infection must be improving on antibiotics. Patients should not require oxygen. Study Chair will be the arbiter of this criterion.

Exclusion Criteria:

1. HIV positive; active hepatitis B or C.
2. Uncontrolled active infections (viral, bacterial, and fungal); the Study Chair will be the final arbiter of this criterion.
3. Patients with active secondary malignancy unless approved by the Study Chair.
4. Liver cirrhosis.
5. Active CNS involvement within the previous 2 months.
6. Prior induction therapy with DAC + CIA.
7. Positive pregnancy test in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization.
8. Breast feeding women.
9. Men must agree not to father a child and agree to use a condom if his partner is of child bearing potential.
10. Inability to comply with medical therapy or follow-up.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2015-09-14 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2021-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Ciurea, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited in MD Anderson Cancer Center
Groups:
- Matched Sibling Donor Group: AML patients with primary induction failure refractory to HD Cytarabine based chemotherapy received matched sibling donor stem cell transplant
- Haploidentical Donor Group: AML patients with primary induction failure refractory to HD Cytarabine based chemotherapy received haplo-identical related donor stem cell transplant
- Matched Unrelated Donor Group: AML patients with primary induction failure refractory to HD Cytarabine based chemotherapy received matched unrelated donor stem cell transplant
Period: Overall Study
Arm/Group | Matched Sibling Donor Group | Haploidentical Donor Group | Matched Unrelated Donor Group
Started | 1 | 8 | 2
Completed | 1 | 6 | 0
Not Completed | 0 | 2 | 2
Not completed — Physician Decision | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Matched Sibling Donor Group | Haploidentical Donor Group | Matched Unrelated Donor Group | Total
Number analyzed (Participants) | 1 | 8 | 2 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 8 | 2 | 11
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 0 | 5
  Male | 0 | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 1 | 7 | 2 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 8 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Overall Response (OR) Post Transplant
Description: Number of participants classified as achieving overall response of complete remission(CR: < 5% blast in a bone marrow/and platelet >100/and ANC >1) or CR without platelet recovery (CRp: < 5% blast in a bone marrow/and platelet <100/and ANC >1) or CR with insufficient hematological recovery (CRi: < 5% blast in a bone marrow/and platelet >100/and ANC <1) post transplant.
Time Frame: 4 months after initial treatment/3 months after transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Sibling Donor Group | Haploidentical Donor Group | Matched Unrelated Donor Group
Number analyzed (Participants) | 1 | 8 | 2
Participants | 1 | 6 | 0

2. Primary Outcome: Treatment-Related Mortality (TRM)
Description: Number of participants died from treatment-related death within 4 months post initial treatment/3 months post transplant.
Time Frame: 4 months post initial treatment/3 months post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Sibling Donor Group | Haploidentical Donor Group | Matched Unrelated Donor Group
Number analyzed (Participants) | 1 | 8 | 2
Participants | 0 | 1 | 0

3. Secondary Outcome: Overall Survival (OS)
Description: Number of participants alive and disease free in 1 year post transplant.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Sibling Donor Group | Haploidentical Donor Group | Matched Unrelated Donor Group
Number analyzed (Participants) | 1 | 6 | 2
Participants | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Matched Sibling Donor Group | Haploidentical Donor Group | Matched Unrelated Donor Group
All-Cause Mortality (participants affected / at risk) | 1/1 | 7/8 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 5/8 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 6/8 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Matched Sibling Donor Group (N=1) | Haploidentical Donor Group (N=8) | Matched Unrelated Donor Group (N=2)
Skin GvHD (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tacrolimus induced PRES (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Secondary Graft Failure due to GvHD (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Fungal Infections (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral Infections (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Matched Sibling Donor Group (N=1) | Haploidentical Donor Group (N=8) | Matched Unrelated Donor Group (N=2)
BK virus associated hemorrhagic cystitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Fluid overload (General disorders) | 1 (1) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 5 (5) | 0 (0)
Mucositis (Gastrointestinal disorders) | 1 (1) | 6 (6) | 0 (0)
Elevated transminitis (Investigations) | 1 (1) | 6 (6) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bacterial Infections (Infections and infestations) | 0 (0) | 6 (6) | 0 (0)
Viral Infections (Infections and infestations) | 0 (0) | 6 (6) | 0 (0)
GI GvHD (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Liver GvHD (Investigations) | 0 (0) | 2 (2) | 0 (0)
Upper GI GvHD (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cytoxan induced cystitis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenic fevers (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Elevated bilirubin (Investigations) | 0 (0) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/03/NCT02441803/Prot_SAP_000.pdf